CLINICAL TRIAL: NCT02530164
Title: Transcranial Direct Current Stimulation (tDCS) As Treatment for Major Depression - A Prospective Multicenter Double Blind Randomized Placebo Controlled Trial (DepressionDC)
Brief Title: Transcranial Direct Current Stimulation (tDCS) As Treatment for Major Depression
Acronym: DepressionDC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Daniel Keeser, Dr. Dipl.-Psych., Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DEP-1483-0152-I
Record Dates: First submitted 2015-08-19; First posted 2015-08-20 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Major Depressive Disorder; Unipolar Depression; Depression
Keywords: tDCS; SSRI; transcranial direct current stimulation; non-invasive brain stimulation; randomized controlled trial; prefrontal tDCS; neuromodulation
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder; Depression | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- real tDCS (Active Comparator)
  Interventions: Device: Transcranial direct current stimulation (tDCS)
- sham tDCS (Placebo Comparator)
  Interventions: Device: Transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Device: Transcranial direct current stimulation (tDCS) — active/sham tDCS as adjunctive treatment with a SSRI

SUMMARY:
Major depressive disorder (MDD) is a common, recurrent, and frequent chronic disorder. Treatment is often challenging; an estimated 20-40% of patients do not benefit sufficiently from existing antidepressant interventions including trials of medication and psychotherapy. A 15-25% of patients manifest a chronic, treatment-resistant course of illness, resulting in a need for additional treatment options. Brain stimulation techniques are considered as a promising therapeutic approach in affective disorders like MDD. Transcranial direct current stimulation (tDCS) is a non-invasive brain stimulation method that has been largely investigated in experimental neurosciences and tDCS of the prefrontal cortex (PFC) has been proposed as novel treatment in MDD. In the largest 2x2 factorial randomized controlled trial in MDD to date, Brunoni et al. (2013) have shown that tDCS combined with an Selective Serotonin Reuptake Inhibitor (SSRI; sertraline) resulted in an antidepressant efficacy superior to placebo treatment, tDCS alone and sertraline alone.

The purpose of this study is to explore the sustained efficacy and tolerability of repeated tDCS for the treatment of MDD. It is hypothesized that prefrontal tDCS in combination with an SSRI will provoke an antidepressant effect while antidepressant medication alone (sham tDCS) did not. This will be measured by the change from baseline in the Montgomery Åsberg Depression Rating Scale (MADRS) scores after 6 weeks of treatment.

In this randomized, placebo-controlled multicenter trial (5 centers involved) patients with a diagnosis of MDD receive a 6-weeks treatment with prefrontal tDCS (anode over electrode position F3, cathode over F4, 5 sessions/week for 4 weeks followed by 2 sessions/week for 2 weeks, 24 treatments in sum, 30min/day, 2mA intensity) or sham tDCS (frequency and duration correspondent active tDCS, ramp in and ramp out periods only without intermittent stimulation), as adjunctive treatment with a SSRI. Follow-up per patient is 3 and 6 months after the last tDCS treatment session. Before, during and after the treatment period different assessment scales will be conducted to record neuropsychological features and the course of the individual symptomatology.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18-65 years of age.
* Primary DSM-5 diagnosis of Major Depression as assessed by the Structured Clinical Interview for DSM-5 Axis I Disorders, Research Version (SCID-5-RV) with a single or recurrent episode with the additional requirements of a current episode with a duration of ≥4 weeks.
* Current depressive episode is less than 5 years duration (the definition of an episode is demarcated by a period of ≥2 months in which the patient did not meet full criteria for the DSM-5 definition of major depressive episode).
* Total HDRS-21 ≥15 at the screening visit.
* The patient did not respond to at least one antidepressant treatment, i.e., a minimum of 1 and a maximum of 4 antidepressant drug trials, of adequate dose and duration (defined as a minimum level of 2 on the ATHF) in the current episode.
* Patient is taking a SSRI of adequate dose and ≥4 weeks (defined as a minimum level of 2 on the ATHF) in the current episode.
* Capable and willing to provide informed consent.
* Negative pregnancy test and willingness to use contraceptive measures during study treatment for women with childbearing potential (i.e <. 2 years post-menopausal)

Exclusion Criteria:

* Investigators, site personnel directly affiliated with this study, and their immediate families (immediate family is defined as a spouse, parent, child or sibling, whether by birth or legal adoption).
* Acute risk for suicide (MADRS, item 10 score of >4 or as assessed by the C-SSRS, agree to item 4 and/or to item 5).
* High degree of therapy resistance defined as >4 sufficient treatment attempts in the current episode (each attempt with an ATHF score of >3).
* Treatment with electroconvulsive therapy in the present episode.
* Treatment with deep brain stimulation or vagus nerve stimulation and/or any other intracranial implants (clips, cochlear implants).
* Any other relevant psychiatric axis-I- and/or axis-II-disorder.
* Any relevant instable medical condition.
* History of treatment with tDCS for any disorder.
* Pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2021-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the Montgomery Åsberg Depression Rating Scale (MADRS) scores at week 6 post-randomization compared to baseline. | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry and Psychotherapy, Ludwig-Maximilian University Munich, Munich, Germany

REFERENCES:
- [Background] Padberg F, Kumpf U, Mansmann U, Palm U, Plewnia C, Langguth B, Zwanzger P, Fallgatter A, Nolden J, Burger M, Keeser D, Rupprecht R, Falkai P, Hasan A, Egert S, Bajbouj M. Prefrontal transcranial direct current stimulation (tDCS) as treatment for major depression: study design and methodology of a multicenter triple blind randomized placebo controlled trial (DepressionDC). Eur Arch Psychiatry Clin Neurosci. 2017 Dec;267(8):751-766. doi: 10.1007/s00406-017-0769-y. Epub 2017 Feb 28. PMID 28246891
- [Derived] Burkhardt G, Kumpf U, Crispin A, Goerigk S, Andre E, Plewnia C, Brendel B, Fallgatter A, Langguth B, Abdelnaim M, Hebel T, Normann C, Frase L, Zwanzger P, Diemer J, Kammer T, Schonfeldt-Lecuona C, Kamp D, Bajbouj M, Behler N, Wilkening A, Nenov-Matt T, Dechantsreiter E, Keeser D, Bulubas L, Palm U, Blankenstein C, Mansmann U, Falkai P, Brunoni AR, Hasan A, Padberg F. Transcranial direct current stimulation as an additional treatment to selective serotonin reuptake inhibitors in adults with major depressive disorder in Germany (DepressionDC): a triple-blind, randomised, sham-controlled, multicentre trial. Lancet. 2023 Aug 12;402(10401):545-554. doi: 10.1016/S0140-6736(23)00640-2. Epub 2023 Jul 3. PMID 37414064
- See also: Related Info — https://www.gcbs.network/gcbs/projects/clinical-trials/Work-Package-7.html